CLINICAL TRIAL: NCT05888792
Title: Myopia Control Effectiveness of Second-generation Defocus Incorporated Multiple Segments Spectacle Lenses on Fast Progressing Myopes: A Randomized Controlled Trial
Brief Title: Myopia Control Efficacy of Second-generation DIMS Spectacle Lenses on Fast Progressing Myopes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: HOYA Lens Thailand LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-ZGET
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: Myopia; Defocus
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either control (wearing single vision lenses) group or treatment (D2 lens) group for first 12 months. After 12 months, the SV lens prescribed to the control group will be replaced with the D2 lens and be monitored for another 12 months. In parallel, the D2 treatment groups will continue their corresponding intervention for 12 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and their guardians will be masked from the grouping. The outcomes assessors will be also masked from the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single vision lens group (No Intervention): Subjects in single vision lens group will receive a pair of single vision lenses for the first year of study. They will then receive a pair of DG2 lenses for the second year of the study.
- D2 lens group (Experimental): Subjects in D2 lens group will receive a pair of D2 lenses over the 2-year study.
  Interventions: Other: Variant of Defocus Incorporated Spectacle lens (DG2)

INTERVENTIONS:
Other: Variant of Defocus Incorporated Spectacle lens (DG2) — DG2 is a variant of Defocus Incorporated Spectacle lens that corrects the distance refraction and provides myopic defocus simultaneously
  Arms: D2 lens group

SUMMARY:
The purpose of this study is to examine the efficacy and performance of the variant of Defocus Incorporated Spectacle lenses on controlling myopia progression in fast progressing myopic children.

DETAILED DESCRIPTION:
The variant of Defocus Incorporated Spectacle lenses (D2) is a multifocal spectacle lens that produces myopic defocus images and corrects distance refractive errors at the same time.

Participants will be randomly allocated to either single vision lens group (control) or the variant of Defocus Incorporated Spectacle lens (D2) group (treatment). After 12 months of lens wear, the SV lens prescribed to the control group will be replaced with the D2 lens and be monitored for another 12 months. In parallel, the D2 treatment groups will continue their corresponding intervention for 12 months. Their cycloplegic refraction and axial length will be monitored every 6 months over 2 years. The changes in refractive errors and axial length in two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* SER: -0.75D or below in both eyes
* Documented history of fast progressing myopia, either in SER or AL

  * SER progression: 0.50D/year or more
  * AL elongation: 0.27mm/year or more
  * For children aged 4-6 years without past prescription forms,
  * 4-5 years old: myopia of -0.75D or below in both eyes
  * 6 years old: myopia of -1.25D or below in at least one eye, with the other eye -0.75D or below
* Best-corrected visual acuity (VA) in both eyes:

  * 4 - 6 years old: 0.20 logMAR (or its equivalent) or better
  * 7-12 years old: 0.00 logMAR (or its equivalent) or better
* Acceptance of random group allocation and the masked study design
* Anisometropia of 1.50 D or less
* Astigmatism of 2.00 D or less

Exclusion Criteria:

* Strabismus and binocular vision abnormalities
* Ocular and systemic abnormalities
* Prior experience of myopia control

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-07-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refraction change in spherical equivalent refraction (SER) | Baseline, 1st year and 2nd year
  Cycloplegic SER (in diopter) will be measured using an open field autorefractor.
  Change in SER with cycloplegia from the baseline over a first 12-month period and a 12-month period of follow-up will be measured

SECONDARY OUTCOMES:
Axial length change | Baseline, 1st year and 2nd year
  Axial length (mm) will be measured after cycloplegia using a non-contact optical biometer.
  Change in axial length from the baseline over a first 12-month period and a 12-month period of follow-up will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yan Yin Tse, PhD, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hon Y, Chun RKM, Leung TW, Qi H, Hasegawa K, Leung KY, To CH, Lam CSY, Tse DY. Myopia control efficacy of second-generation defocus incorporated multiple segments spectacle lenses on fast progressing myopes: Study protocol of a randomised controlled trial. PLoS One. 2025 Oct 31;20(10):e0335061. doi: 10.1371/journal.pone.0335061. eCollection 2025. PMID 41171741